CLINICAL TRIAL: NCT06565494
Title: A Pilot Study of Midomafetamine (MDMA-Assisted) Therapy for the Treatment of Pathological Narcissism
Brief Title: MDMA-Assisted Therapy for Pathological Narcissism
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Anthony Back MD, Professor, Department of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020440
Record Dates: First submitted 2024-07-26; First posted 2024-08-22 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Narcissism
Keywords: MDMA; Assisted Therapy; midomafetamine
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Open-Label, proof-of-concept with single group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participant (Experimental): midomafetamine (MDMA)-assisted therapy
  Interventions: Drug: midomafetamine (MDMA)-Assisted Therapy

INTERVENTIONS:
Drug: midomafetamine (MDMA)-Assisted Therapy — This treatment consists 3 Preparation sessions followed by 3 Experimental sessions at 4-week intervals; after each Experimental session, 3 weekly Integration sessions will be conducted. For the first Experimental Session, the dose of MDMA is 80 mg; for the second and third Experimental Sessions, the dose of MDMA is 120 mg. For all three Experimental sessions, a supplemental dose of 50% of the initial dose will be available. The Preparation, Experimental, and Integration Sessions will involve psychotherapy developed specifically for this trial and population.

SUMMARY:
This open-label, proof-of-concept pilot study will assess the efficacy and safety of midomafetamine (MDMA) - assisted therapy (AT) for participants diagnosed with pathological narcissism. As all participants will be allocated to a single group assignment, there will be no blinding, randomization, or comparator treatment. Participants will have a screening visit, a preparation period of 3 visits, a treatment period receiving MDMA-AT at 3 monthly visits, a 6 month follow up period coming in at one week, one month, three months and six months after last treatment visit.

DETAILED DESCRIPTION:
This open-label, proof-of-concept pilot study will assess the efficacy and safety of midomafetamine- assisted therapy (MDMA-AT) for participants diagnosed with pathological narcissism. As all participants will be allocated to a single group assignment, there will be no blinding, randomization, or comparator treatment.

Up to 12 participants will be enrolled. Each participant will have 2 informants, one family member and one psychotherapist.

The visit schedule for each participant will be comprised of the following:

* Screening Period: phone screen, visit screen, informed consent, eligibility assessment, and enrollment invitation to eligible participants;
* Preparation Period: medication tapering, three Preparation Sessions, Baseline assessments, Enrollment Confirmation;
* Treatment Period: three monthly Experimental Sessions and nine associated Integration Sessions over ~12 weeks;
* Follow-up Period and Study Termination: four Follow-up Visits at one week, one month, three months and six months after the final Integration Session to collect clinical outcome measures; Study Termination will happen at the last Follow-up Visit.

The treatment (MDMA-AT) consists 3 Preparation sessions followed by 3 Experimental sessions at 4-week intervals; after each Experimental session, 3 weekly Integration sessions will be conducted. For the first Experimental Session, the dose of MDMA is 80 mg; for the second and third Experimental Sessions, the dose of MDMA is 120 mg. For all three Experimental sessions, a supplemental dose of 50% of the initial dose will be available. The Preparation, Experimental, and Integration Sessions will involve psychotherapy developed specifically for this trial and population.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years old.
2. Are between the ages of 18 years old and 64 years old.
3. Weigh at least 48 kilograms (i.e., 106 pounds).
4. If able to become pregnant, must have a negative over-the-counter (OTC) urine pregnancy test at the Screening Visit, at the last Preparation Session, and prior to each Experimental Session. They must agree to use adequate birth control from Enrollment Confirmation through 10 days after the last Experimental Session. Adequate birth control methods include intrauterine device (IUD), injected, implanted, intravaginal, or transdermal hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e., condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom). "Not able to become pregnant" is defined as permanent sterilization, postmenopausal (defined as 12 months with no menses without an alternative medical cause), or assigned male at birth. All subjects who do not fall into the category of 'not able to become pregnant' will complete pregnancy tests immediately before every Experimental Dosing Session.
5. If assigned male at birth, must agree to use barrier contraception if partner is of childbearing potential, and must agree to consider sperm donation if planning to conceive after completing study participation.
6. Are proficient in speaking and reading English.
7. Are able to give adequate informed consent.
8. Are able to swallow pills.
9. Must agree to safety lab assessments including a complete blood count and a metabolic panel inclusive of kidney and liver function tests.
10. Must agree to a screening 12-lead ECG that is evaluated by a qualified cardiologist to rule out any baseline cardiac abnormalities which would lead to enrollment exclusion; if a 12-lead ECG has been obtained in the last 12 months that has been evaluated by a qualified cardiologist, this may be used for screening purposes in which case participants must sign a medical release in order for study investigators to obtain a copy for review.
11. Must agree to a 1-minute rhythm strip at the Screening Visit to assess for heretofore undiagnosed arrhythmias.
12. Must agree to commit to the midomafetamine (MDMA) dosing, Experimental Sessions, non-drug Preparation and Integration Sessions, Follow-up Visits to complete clinical measures at all four Follow-up endpoints, and all necessary telephone contact.
13. Must select a family member (spouse/partner or relative) with whom they are willing to allow Study Staff to communicate and whom they consent to complete Informant-report assessments at Baseline (T0) and at all Follow-up endpoints (T1-T4). Contact information (cell phone & email address) for their selected family member must be provided by participant at the Screening Visit. Participant's selected family member must consent to participate and provide written informed consent.
14. Must be willing to sign a medical release for Study Staff to communicate directly with the participant's psychotherapist and consent to their completing Informant-report assessments at Baseline (T0) and at all Follow-up intervals (T1-T4). Contact information (business and/or cell phone) for their psychotherapist will be provided by participant at the Screening Visit. Participant's psychotherapist must consent to participate and provide written informed consent.
15. Must provide a contact (spouse/partner, relative, close friend, or other caregiver) who is willing and able to be reached by Study Staff in the event of an emergency, if the participant becomes suicidal, or if the participant is unreachable.
16. Must agree to inform the Study Staff within 48 hours if any medical conditions occur or medical procedures are planned.
17. Must agree not to participate in any other interventional clinical trials during the duration of this study without prior approval of the study investigators.
18. Must avoid starting any new prescription medications (with the exception of contraception medications, thyroid hormones, or other medications approved by the study investigators).
19. Are willing to comply with all medication requirements per protocol.
20. Must be willing to taper off all prohibited medications and substances with drug-drug interactions with MDMA for at least five half-lives of the drug plus one week for stabilization to ensure an appropriate medication washout to avoid the possibility of interactions prior to the third Preparation Session. Must also agree not to resume any prohibited non-psychoactive medications until 40 hours (five half-lives of MDMA) after the last Experimental Session. Must agree to sign a medical release for Study Staff to communicate with the participant's prescribing physician who will direct medication tapers.
21. Must be willing to taper off all prohibited psychoactive medications (including SSRIs, SNRIs, MAOIs, other antidepressants) as well as other psychoactive medications (including mood stabilizers and anti-psychotics) and psychoactive substances to ensure an appropriate washout prior to the third Preparation Session when Baseline outcome measures are obtained. Must also agree not to resume any of these medications until all primary outcome data is collected at the time of Study Termination unless restarting is required/or in the best interest of the participant. Must agree to sign a medical release for Study Staff to communicate with the participant's prescribing physician who will direct medication tapers.
22. Must be willing to work with their outside prescribing physician(s) who will direct and oversee the tapering of all prohibited medications.
23. Are able to decrease dose of allowable opiates, if used for pain management, leading up to the Experimental Session in order to avoid taking the medication prior to the initial MDMA administration and 24 hours after. During this period, the participant will be allowed to take the medication if needed for intolerable pain flare-ups or to prevent withdrawal symptoms.
24. Agree to attending all the study sessions, and agree not to be enrolled on another interventional clinical trial without approval of the study investigators for the duration of this study.
25. Are willing to attend Experimental and Integration Sessions without a support-person present; while some previous trials have permitted support persons to be present for portions of the Treatment Period, the presence of a family member may inhibit patients with pathological narcissism who struggle with shame and fear of exposure.
26. Must arrange for transportation after each Experimental Session and for travel the following day to-and-fro the first Integration Session.
27. Must agree not to operate a vehicle for at least 24 hours after the dosing of each Experimental Session.

    Psychiatric Conditions
28. At the Screening Visit, must meet criteria for a diagnosis of pathological narcissism per the Diagnostic and Statistical Manual of Mental Disorders - 5th edition (DSM-5) Section III Alternative Model for Personality Disorders (AMPD). (Prior to invitation to the Screening Visit, all participants will have been pre-screened with questions from the Personality Diagnostic Questionnaire - Version 4+ (PDQ-4+) to assess for the DSM-IV/5 Section II diagnostic criteria for NPD and the Super Brief Pathological Narcissism Inventory (SB-PNI) to assess for narcissistic grandiosity and narcissistic vulnerability consistent with pathological narcissism.)
29. Must be in an ongoing (greater than 6 months) outpatient individual psychotherapy with a clinically licensed psychotherapist who agrees the participant's primary diagnosis is pathological narcissism. Need to be known to their psychotherapist for at least six months or to the study team as a patient of Dr. Albert for at least six months.
30. Must agree to continue their ongoing psychotherapy with their psychotherapist through the 12-week Treatment Period.

    Medical Conditions
31. May have well-controlled hypertension that has been successfully treated with anti-hypertensive medicines.
32. May have asymptomatic Hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed.
33. May have a history of or current Diabetes Mellitus if screening rules out cardiovascular disease that would meet an exclusion criterion and the condition is judged to be stable on effective management.
34. May have hypothyroidism if taking adequate and stable thyroid replacement medication.
35. May have a history of or current glaucoma if approval for study participation is received from an ophthalmologist.
36. If there are any questions about possible medical problems, the study physician will request additional tests, assessments, or measures as indicated. The study physician may also contact outside providers with participant permission as needed.
37. Additional visits (in person, by telephone, or via telemedicine) may be scheduled at the discretion of the study investigators to collect more information for determining eligibility or to discuss study expectations with the potential participant.

Exclusion Criteria:

1. Are not able to give adequate informed consent.
2. Are less than 18 years old or 65 years or older.
3. Have any current problem which in the opinion of the study investigators, study physician or Medical Monitor might interfere with participation including:

   Psychiatric Conditions
4. Have a psychiatric diagnosis of bipolar disorder, psychotic disorder, anorexia nervosa or bulimia as assessed with the Mini International Neuropsychiatric Interview (MINI) at the Screening Visit.
5. Have had active suicidal ideation and/or behaviors in Past 12 Months as assessed with the MINI at the Screening Visit. For those assessed to be at Moderate Risk or High Risk "likely in the near future" using the established MINI thresholds, participants' personal therapists will be contacted to assist in triage planning. If it is determined that the participant is at imminent risk of suicide and/or the personal therapist is unavailable, emergency services will be called for transfer to the nearest Emergency Department and "a "warm hand-off" will be made to a receiving provider there.
6. Have a current alcohol or substance use disorder as assessed with the MINI at the Screening Visit.
7. Have a co-occurring dissociative identity disorder diagnosis from their current clinically licensed psychotherapist.
8. Have used MDMA within the last 12 months.

   Medical Conditions
9. Have uncontrolled hypertension using the standard criteria of the American Heart Association (values of 140/90 milligrams of Mercury [mmHg] or higher assessed on three separate occasions).
10. Have a history of ventricular arrhythmia at any time, other than occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease. Have a history of atrial flutter or any arrhythmia at any time, other than occasional PVCs in the absence of ischemic heart disease. Participants with a history of paroxysmal supraventricular tachycardia, paroxysmal atrial tachycardia, or atrial fibrillation arrhythmia may be enrolled if successfully treated with ablation cardioversion treatment at least 12 months prior and cleared by a cardiologist, the site physician, and Medical Monitor.
11. Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
12. Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds corrected by Bazett's formula).
13. Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
14. Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate. This includes, but is not limited to, a history of myocardial infarction, angina that meets criteria for Canadian cardiovascular class II, III, or IV, cerebrovascular accident, or aneurysm. Participants with other mild, stable chronic medical problems may be enrolled if the study investigators, study physician, and Medical Monitor agree the condition would not significantly increase the risk of MDMA administration or be likely to produce significant symptoms during the study that could interfere with study participation or be confused with side effects of the IMP.
15. Have symptomatic liver disease with liver function tests (AST/ALT/ALP) 1.5x greater than the upper limits of normal.
16. Have history of hyponatremia or hyperthermia.
17. Weigh less than 48 kilograms (kg).
18. Are pregnant or lactating or nursing, or are of childbearing potential and are not practicing an adequate birth control method. Adequate birth control methods include intrauterine devices (IUD), injected, implanted, intravaginal, or transdermal hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Narcissism Inventory (PNI)--Participant version | Baseline, After each MDMA session (approx every month for 3 months); After MDMA sessions end, 1 month, 3 months, 6 months
  Assess changes in diagnostic features of pathological narcissism per self-report. This measure has 52 items each rated on a 6-point Likert scale with higher scores indicating higher severity.

OTHER OUTCOMES:
Reported adverse events | Baseline, After each MDMA session (approx every month for 3 months); After MDMA sessions end, 1 month, 3 months, 6 months
  Assess incidence of adverse events that may be indicative of an acute medical complication of MDMA, for example, chest pain, shortness of breath, or neurological symptoms or any other signs or symptoms that prompt additional vital sign measurements. Assess incidence of AEs by severity and by severity categorized as leading to discontinuation of MDMA, resulting in death or hospitalization, or continuing at Study Termination. Assess incidence of Treatment Emergent AEs (TEAEs) to determine relationship to the MDMA based on relative incidence. Assess incidence of TEAEs by severity reported during an Experimental Session, 1 day, and 2 days after each Experimental Session.
Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline, After each MDMA session (approx every month for 3 months); After MDMA sessions end, 1 month, 3 months, 6 months
  Assess incidence of positive or serious ideation and suicidal behavior. The screening version of this measure produces a 'low', 'moderate', or 'high' risk of suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Back, MD, Principal Investigator — University of Washington; Alexa Albert, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This website contains information for anyone who is interested in learning more or participating in the study. — https://depts.washington.edu/mdma-narcissism/